CLINICAL TRIAL: NCT01180244
Title: The Clinical Effect of Low-Intensity Electromagnetic Field Neurostimulation in Fibromyalgia Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McLaren Regional Medical Center (Other)
Collaborators: Kettering University (Other)
Responsible Party: Principal Investigator, Jeffrey B. Hargrove, Principal Investigator, McLaren Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; noninvasive; electrical; cortical; stimulation; pain; brain; tender point
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Active Comparator): Subjects in this group will receive the noninvasive cortical stimulation signal from the treatment device
  Interventions: Device: Noninvasive cortical electrical stimulation
- Placebo group (Placebo Comparator): Subjects in this group will be provided the same experience as those in the active treatment arm, but will not receive the noninvasive cortical stimulation signal from the treatment device
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Noninvasive cortical electrical stimulation — Subjects will receive 22 sessions of the intervention protocol, twice per week for a total of 11 weeks. The signal stimulation used in this study utilizes amplitude modulation to shape a high frequency carrier signal, nominally greater than 10 kilohertz, into the form of one or more low frequency components, nominally less than 40 hertz. Exact protocol is set in software and is the same for all participants in the active treatment arm.
  Other Names: NeuroPoint
  Arms: Active treatment
Device: Sham treatment — Subjects in the placebo group will receive the exact same experience as those in the active treatment group. However, the device will not output any electrical stimulation signal.
  Other Names: NeuroPoint
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine whether persons treated with a low-intensity, noninvasive form of cortical electrical stimulation experience a reduction in symptoms of fibromyalgia different than persons receiving a sham treatment. Outcome measures include reduction in patient pain levels and improvement in sleep measures.

DETAILED DESCRIPTION:
There is increasing acceptance that pain in fibromyalgia is a result of dysfunctional sensory processing in the spinal cord and brain. Electrical cortical stimulation is a device-based form of therapy that is increasingly being considered as an adjuvant to current medical modalities for the treatment of chronic pain conditions such as fibromyalgia. The investigators propose that stimulation of cortical areas believed to be involved in dysfunctional sensory processing may have a beneficial influence on fibromyalgia symptoms.

The aim of this randomized double blind, placebo controlled study is to evaluate the efficacy, safety, and tolerability of noninvasive cortical stimulation in the management of fibromyalgia symptoms. More specifically, an active treatment group of subjects will receive the study's cortical stimulation protocol twice a week for 11 weeks and will be evaluated within 14 days following end of treatment, for a total timeframe of 13 weeks. In comparison, a similar group of subjects will receive the same treatment protocol without the actual stimulation signal being applied. The signal utilized is a modulated form that permits very low-intensity signals to pass through outer tissues with less attenuation due to tissue impedance. The signals are of a sufficiently low strength that they are below the level of perception. Hence subjects cannot feel the signal, and are therefore blinded to treatment arm. Investigators and clinical staff are also blinded. Outcome measures include post-treatment to baseline changes in tender points, sleep characteristics as measured by visual analog scales, and outcomes instruments including the Fibromyalgia Impact Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 65 years
* An ability to read and comprehend English
* Completion of a minimum of grade 8 education
* Diagnosis of fibromyalgia in 1999 or earlier, by a rheumatologist or appropriate specialist, and currently meeting the American College of Rheumatology 1990 criteria
* Symptoms for at least 48 months with no recent remission of symptoms to any degree

Exclusion Criteria:

* Developmental disabilities, or significant psychological disorder (except depression and anxiety disorders) for which treatment has become necessary
* A history of chronic infection or chronic condition such as lupus, rheumatoid arthritis, Parkinson's Disease, multiple sclerosis, hepatitis, history of meningo-encephalitis, polio, seizures, or metastatic cancer
* Current pregnancy, or plans to become pregnant during the study period.
* Any other condition deemed to pose a risk to the patient at the discretion of the investigators
* Exposure to other neurostimulation systems, or electroconvulsive therapy
* Any implantable electronic device
* Any present or previous litigation regarding their physical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2002-01; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Hargrove, PhD, Principal Investigator — Kettering University; Susan J Smith, MD, Principal Investigator — McLaren Regional Medical Center; Sunil Nagpal, MD, Principal Investigator — McLaren Regional Medical Center; David G Simons, MD, Principal Investigator — Emory University
Locations (1):
- McLaren Regional Medical Center, Flint, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo Group
Started | 45 (Number of enrolled patients initially randomized to active treatment group) | 46 (Number of enrolled patients initially randomized to placebo group)
Received Treatment | 40 (Number of patients in the active treatment group that received at least one study treatment) | 45 (Number of patients in the placebo group that received at least one sham treatment)
Completed | 39 (Number of active treatment patients who completed all study visits and are evaluable) | 38 (Number of placebo group patients who completed all study visits and are evaluable)
Not Completed | 6 | 8
Not completed — Lack of Efficacy | 0 | 7
Not completed — Physician Decision | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Group | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.3) | 54.0 (9.0) | 52.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 71
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change in Tender Point Pain Threshold
Description: Tender point pain threshold is derived by summing the dolorimetry-based pain pressure thresholds measured on a subject for each of the 18 tender points sites specified by the American College of Rheumatology for fibromyalgia classification. The range of dolorimeter values for each tender point site is 0-4 (units are kilograms per square centimeter, i.e. kg/cm^2). Higher numbers represent greater pressure required to elicit pain, and are thus indicators of "less pain" sensitivity at the tender point. Since 18 tender points are measured on a patient and their individual dolorimeter values summed, the range of tender point pain threshold values is 0-72. A higher score represents less overall pain sensitivity. The change in tender point pain threshold is determined by subtracting values at baseline from values at end of treatment. Thus a positive difference represents pain improvement (i.e.. a better outcome). A negative difference represents pain worsening (i.e. a worse outcome).
Time Frame: Total timeframe 13 weeks: baseline followed by 11 weeks of treatment with outcome assessed within 14 days following end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment | Placebo Group
Number analyzed (Participants) | 39 | 38
units on a scale | 19.6 (8.4) | -3.2 (9.4)

2. Secondary Outcome: Change in Number of Positive Tender Points
Description: The number of positive tender points ranges from 0-18, and are defined per criteria set forth by the American College of Rheumatology and based on dolorimetry measurements made on 18 prescribed tender point locations. A tender point is considered "positive" if less than 4 kilograms per centimeter squared pressure is required to elicit a painful response. The change in number of positive tender points is determined by subtracting the number of positive tender points at baseline from the number of positive tender points at end of treatment. Thus, a negative number represents pain improvement (i.e. better outcome), whereas a positive number represents a worsening of pain (i.e. worse outcome).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of positive tender points
Arm/Group | Active Treatment | Placebo Group
Number analyzed (Participants) | 39 | 38
Number of positive tender points | -7.4 (4.4) | -0.2 (2.3)

3. Secondary Outcome: Change in Fibromyalgia Impact Questionnaire Overall Score
Description: The Fibromyalgia Impact Questionnaire yields a score ranging from 0 to 100, with higher scores representing a greater impact or level of symptoms. The change in Fibromyalgia Impact Questionnaire is determined by subtracting scores at baseline from scores at end of treatment. Thus negative numbers represent symptom improvement (i.e. a better outcome) and positive numbers represent symptom worsening (i.e. a worse outcome).
Time Frame: as for outcome 1
Population: Participants who correctly completed the outcome questionniare
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment | Placebo Group
Number analyzed (Participants) | 36 | 35
units on a scale | -15.5 (20.2) | -5.6 (16.4)

4. Secondary Outcome: Change in Fibromyalgia Impact Questionnaire Pain Visual Analog Scale
Description: The Fibromyalgia Impact Questionnaire includes a pain visual analog scale (VAS) with ranges of 0-10 centimeters. Higher values represent greater pain. The change in Fibromyalgia Impact Questionnaire pain visual analog scale is determined by subtracting baseline VAS values from end of treatment VAS values. Thus, a negative value represents pain improvement (i.e. a better outcome), while a positive value represents pain worsening (i.e. a worse outcome).
Time Frame: as for outcome 1
Population: Participants who correctly completed the outcome questionniare
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment | Placebo Group
Number analyzed (Participants) | 36 | 35
units on a scale | -2.0 (3.0) | -0.6 (2.5)

5. Secondary Outcome: Change in Fibromyalgia Impact Questionnaire Sleep Satisfaction Visual Analog Scale
Description: The Fibromyalgia Impact Questionnaire includes a sleep visual analog scale (VAS) with ranges of 0-10 centimeters. Higher values represent greater difficulty with sleep. The change in Fibromyalgia Impact Questionnaire sleep visual analog scale is determined by subtracting baseline VAS values from end of treatment VAS values. Thus, a negative value represents sleep improvement (i.e. a better outcome), while a positive value represents sleep worsening (i.e. a worse outcome).
Time Frame: as for outcome 1
Population: Participants who correctly completed the outcome questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment | Placebo Group
Number analyzed (Participants) | 36 | 35
units on a scale | -2.1 (2.5) | -0.7 (2.4)

ADVERSE EVENTS:
Time Frame: Total timeframe 13 weeks: 11 weeks of treatment with outcome assessed within 14 days following end of treatment
Arm/Group | Active Treatment | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 0/45 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes